CLINICAL TRIAL: NCT05287178
Title: Integration of DBT Skills and Parent Training for Parents With a History of Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00000041; P50DA048756 (NIH)
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2022-03

CONDITIONS: Parenting; Substance Abuse Relapse; Emotional Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBT Skills + Parent Training (Experimental): The DBT Skills +PT group intervention integrates DBT Skills, Parent Management Training (PMT), and Emotion Coaching (EC). Each session includes a mindfulness practice, homework review to discuss use of skills previously learned, didactics to learn a new set of DBT and PT skills, and assignment of homework. The DBT Skills portions cover the four modules of traditional DBT Skills: Mindfulness, Emotion Regulation, Distress Tolerance (including skills specifically focused on managing difficulties with addiction), and Interpersonal Effectiveness. PT skills include both PMT and EC components such as: praise, use of parental attention to reward positive behavior, reward systems, effective commands and consequences, psychoeducation on children's emotional development, teaching children to label emotions, validating children's emotions, and handling children's negative emotions, and fostering positive emotions.
  Interventions: Behavioral: DBT Skills + Parent Training

INTERVENTIONS:
Behavioral: DBT Skills + Parent Training — The DBT Skills +PT group intervention integrates DBT Skills, Parent Management Training (PMT), and Emotion Coaching (EC). Each session includes a mindfulness practice, homework review to discuss use of skills previously learned, didactics to learn a new set of DBT and PT skills, and assignment of homework. The DBT Skills portions cover the four modules of traditional DBT Skills: Mindfulness, Emotion Regulation, Distress Tolerance (including skills specifically focused on managing difficulties with addiction), and Interpersonal Effectiveness. PT skills include both PMT and EC components such as: praise, use of parental attention to reward positive behavior, reward systems, effective commands and consequences, psychoeducation on children's emotional development, teaching children to label emotions, validating children's emotions, and handling children's negative emotions, and fostering positive emotions.

SUMMARY:
This treatment development study is aimed at developing and pilot testing a 20-week remotely delivered group intervention that integrates two evidence-based treatments: 1) Dialectical Behavior Therapy (DBT) Skills - targeting parental emotion dysregulation and substance use, and 2) Parent Training (PT) - targeting parenting behaviors linked to children's mental health. The case study will provide preliminary data on the feasibility of the DBT Skills +PT intervention and its engagement of the targeted outcomes, and aims to complete foundational steps necessary to conducting a future, larger scale randomized controlled trial.

Specific aims are to:

1. Determine feasibility, acceptability and implementation.
2. Evaluate pre-post changes in measures of parental emotion dysregulation, parenting quality and children's mental health.

DETAILED DESCRIPTION:
Overview

This treatment development study is aimed at developing and pilot testing a 20-week remotely delivered group intervention that integrates two evidence-based treatments: 1) Dialectical Behavior Therapy (DBT) Skills - targeting parental emotion dysregulation and substance use, and 2) Parent Training (PT) - targeting parenting behaviors linked to children's mental health. The case study will provide preliminary data on the feasibility of the DBT Skills +PT intervention and its engagement of the targeted outcomes, and aims to complete foundational steps necessary to conducting a future, larger scale randomized controlled trial. Specific aims are to:

1. Determine feasibility, acceptability and implementation. Number of sessions attended by parents and attrition rates will be assessed to determine overall feasibility of the intervention. Acceptability will be evaluated using measures of client satisfaction. Implementation will be assessed by examining the frequency with which clients report using DBT and parenting skills.
2. Evaluate pre-post changes in measures of parental emotion dysregulation, parenting quality and children's mental health. Across 12 parents (three groups with ~4 parents in each group), we will evaluate the change in these interlinked domains which represent risk factors for relapse and further adverse outcomes. We anticipate pre-post changes (2 time points, approximately 20-22 weeks apart) will be comparable to well-established change scores from the clinical trial literature base for DBT Skills and parent training interventions.

The study will be conducted remotely and involves five phases: 1) an online screener questionnaire; 2) a clinical diagnostic intake interview to formally determine eligibility; 3) an online pre-intervention assessment survey; 4) 20 weeks of DBT Skills +PT group therapy; 5) an online post-intervention assessment survey. All online screeners and assessments will be completed using Qualtrics. The clinical diagnostic intake interview, weekly DBT Skills +PT sessions and exit interviews will all be conducted over a HIPAA compliant version of Zoom.

Assignment of Participants to Condition All participating parents will be assigned to the DBT Skills +PT condition. Up to 12 parents will be enrolled in the DBT Skills +PT group therapy. As the intervention is scheduled for 20 weeks, families will be recruited twice throughout the year to facilitate running 3 groups (~4 participants in each).

Data Analysis Results from this case study to pilot test the integrated DBT Skills +PT intervention will be descriptive. For Aim 1, feasibility of the intervention will be evaluated by calculating the average number of sessions attended by parents and attrition rates. Acceptability will be examined by averaging the total scores obtained from the Client Satisfaction Questionnaire (CSQ-8). We will examine implementation by calculating the average daily number of DBT and parenting skills parents report using each week on their diary card (averaged across parents) and comparing these to skill use reported in other published research. We will primarily report data for Aim 1 at an aggregated group level.

For Aim 2, we will examine pre-post changes for primary and secondary outcomes - parental emotion dysregulation, parenting quality, child internalizing and externalizing behaviors, child emotion regulation, and parent mental health symptoms. Pre-post change scores will be compared to the clinical trial literature base for DBT and parent training interventions which often use the same measures and for which expected change scores are established.

ELIGIBILITY:
Inclusion Criteria:

Participants must reside in Oregon.

Participants must have at least partial custody of a preschool-aged child (3-6 years)

Participants must present elevated levels of emotion dysregulation on the Difficulties with Emotion Regulation Scale (DERS) (a score of >88, equivalent to +.5 SD above a normative score) on the online screener.

Participants must endorse 2 or more positive answers on adapted version of the CAGE-AID screener for drug and alcohol problems, which asks about substance use in the past 5 years.

Participants must meet diagnostic criteria for a past (past 5 years) but not current (past 12 months) substance use disorder (SUD) from the following DSM 5 defined disorders: alcohol, cannabis, hallucinogenic, inhalant, opioid, sedative/hypnotic/anxiolytic, and stimulant.

Participants must be proficient in English.

Participants must have the internet access needed to participate in an online remote telehealth intervention.

Exclusion Criteria:

Participants will be excluded if they or their child have a known developmental disability or if during the clinical intake parents are determined to have a low IQ score (IQ<70) on the PPVT-V.

Participants will be excluded if they are psychotic as determined by the SCID 5.

Participants will be excluded if they are actively manic or psychotic as determined by clinical observation.

Participants will be excluded if they are actively suicidal with an active plan as determined by the SCID 5 and/or Patient Health Questionnaire 9 (PHQ-9).

Participants will be excluded if they are determined by clinical judgment to be at high risk of violence towards others.

Participants may be excluded if clinical judgment suggests they requires a higher level or different form of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon, Eugene, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parents were recruited via a variety of methods (e.g. university departmental database; social media; Craigslist; community mental health referrals; direct mailing through Early Head Start). Parents were recruited multiple times throughout the year to facilitate running three groups. Group 1 sessions ran from July until December 2021. Groups 2 and 3 ran from March 2022 until August 2022.
Pre-assignment Details: Of 17 participants who consented, 13 met eligibility criteria. One chose not to participate and 12 were enrolled in the DBT Skills + Parent Training intervention.
Groups:
- DBT Skills + Parent Training: The DBT Skills +PT group intervention integrates DBT Skills, Parent Management Training (PMT), and Emotion Coaching (EC).
Period: Overall Study
Arm/Group | DBT Skills + Parent Training
Started | 12
Completed | 10
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.75 (6.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Difficulties with Emotion Regulation Scale (DERS) [Mean (Standard Deviation); unit: units on a scale] — Used in this study as a measure of parental emotion dysregulation. The DERS is a 36-item self-report measure used to assess adult emotion dysregulation. Items are rated on a scale of 1 to 5, and total scores range from 36 to 180, with higher scores indicating higher levels of dysregulation.
  units on a scale | 109.50 (13.33)

OUTCOME MEASURES:

1. Primary Outcome: Parental Emotion Dysregulation - The Difficulties With Emotion Regulation Scale (DERS)
Description: The Difficulties with Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) is a 36-item self-report measure used to assess adult emotion dysregulation. Items are rated on a scale of 1 to 5, and total scores range from 36 to 180, with higher scores indicating higher levels of dysregulation.
Time Frame: Baseline and post-intervention (22 week timepoint)
Population: 2 participants lost to post-intervention follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 12
units on a scale
  Baseline | 109.50 (13.33)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 68.80 (28.88)

2. Primary Outcome: Parenting Stress - Parenting Stress Index Short Form
Description: The Parenting Stress Index Short Form (PSI-4 SF; Abidin, 1995) is a 36-item parent report measure of parental stress (rated on a five point Likert scale), and includes three subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Raw Subscale scores are summed into a Total Stress score that ranges from 36 to 180, with higher scores indicating higher levels of parenting stress. Normative scores have been established and raw scores are then converted to percentiles for interpretation.
Time Frame: Baseline and post-intervention (22 week timepoint)
Population: 2 participants lost to post-intervention follow-up
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 12
percentile
  Baseline | 68.92 (16.71)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 48.00 (24.33)

3. Primary Outcome: Parenting Quality (Total Dysfunctional Discipline) - The Parenting Scale
Description: The Parenting Scale (PS; Arnold et al., 1993) is a 30-item self-report questionnaire, in which parents are asked to describe (on a Likert scale of 1-7) how they respond to a variety of child misbehaviors. In addition to three sub scales (laxness, over-reactivity and hostile parenting), it yields a total dysfunctional discipline score, which is calculated by averaging responses on all items. Total scores can thus range from 1 to 7, with higher scores reflecting greater dysfunctional discipline.
Time Frame: Baseline and post-intervention (22 week timepoint)
Population: 2 participants lost to post-intervention follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 12
score on a scale
  Baseline | 3.62 (.51)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 2.75 (.81)

4. Primary Outcome: Parental Emotion Socialization (Non-supportive Parenting) - Coping With Children's Negative Emotions Scale (CCNES)
Description: The Coping with Children's Negative Emotions Scale (CCNES; Fabes, Eisenberg & Bernzweig, 1990) assesses parental self-report of emotion socialization practices. Parents are presented with 12 vignettes describing scenarios in which their children exhibit distress. Parents rate (on a Likert scale of 1-7) the likelihood they would engage in 6 potential parental responses to these situations, with each corresponding to 6 subscales which are each mean-scored: distress reactions, punitive reactions, minimization, expressive encouragement, emotion-focused reactions and problem-focused reactions. The first three can then be summed and mean-scored into an Invalidating/non-supportive composite and the latter three can be summed and mean-scored into a Validating/Supportive composite. Scores for the composites range from 1 to 7 with higher scores indicating higher levels of non-supportive or supportive parenting.
Time Frame: Baseline and post-intervention (22 week timepoint)
Population: 2 participants were lost to follow up/post-intervention assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 12
score on a scale
  Baseline | 2.43 (.62)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 2.16 (.60)

5. Primary Outcome: Acceptability (Client Satisfaction) - Client Satisfaction Questionnaire (CSQ-8)
Description: The Client Satisfaction Questionnaire (CSQ-8; Attkisson & Zwick, 1982) will be used to assess acceptability of the intervention. It is a brief 8-item self-report measure in which clients are asked to rate (on a Likert scale of 1-4) their satisfaction with the intervention. Scores range from 8 to 32 with higher scores indicating greater satisfaction.
Time Frame: Post-intervention (22 week timepoint)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 8
score on a scale | 30.75 (2.82)

6. Primary Outcome: Feasibility of Intervention (Attendance)
Description: Average number of sessions attended
Time Frame: Post-intervention (20 week timepoint)
Population: Treatment completers
Measure: Mean (Standard Deviation); unit: percentage of sessions attended
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 8
percentage of sessions attended | 86.25 (15.75)

7. Primary Outcome: Feasibility of Intervention (Attrition)
Description: Attrition rate was measured as percentage of participants who discontinued treatment.
Time Frame: Post-intervention (20 week timepoint)
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 12
Participants | 4

8. Primary Outcome: Implementation of Skills
Description: Weekly avg. number of DBT and parenting skills used daily
Time Frame: Baseline up to 22 weeks
Population: Treatment completers who completed weekly daily diaries on skill use
Measure: Mean (Standard Deviation); unit: number of skills used daily
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 7
number of skills used daily
  DBT Skills in non-parenting contexts | 2.56 (2.32)
  DBT Skills in parenting contexts | 1.53 (1.85)
  Parent Training skills | 4.03 (3.65)

9. Secondary Outcome: Child Externalizing Behaviors - Child Behavior Checklist (CBCL)
Description: The Child Behavior Checklist (CBCL; Achenbach & Rescorla, 2000) is a 99-item parent-report ratings scale (items are rated from 0-2) for children's problem behaviors. The scale provide subscales for both internalizing (e.g. anxious, sad) and externalizing (e.g. hyperactive, aggressive) behaviors. Normative scores have been established and total summed raw scores are converted to T-scores and percentiles for interpretation. T-scores range from 28 to 100, with a population mean of 50 and a standard deviation of 10. Higher T-scores indicate greater problem behaviors and symptoms of psychopathology.
Time Frame: Baseline and Post-intervention (22 week timepoint)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 10
T-score
  Baseline | 53.00 (9.87)
  Post-intervention | 44.90 (10.71)

10. Secondary Outcome: Child Emotion Dysregulation - Emotion Regulation Checklist (Lability/Negativity Subscale)
Description: The Emotion Regulation Checklist (ERC; Shields & Cicchetti, 1997) is a 24-item parent-report measure in which parents rate (on a Likert scale of 1-4) how characteristic of their child are statements which focus on mood lability, lack of flexibility, dysregulated negative emotion, empathy, emotional self-awareness and positive response to others. Items are summed to produce produce two subscales (lability/negativity and emotion regulation). The negativity/lability subscale ranges from 15 to 60 with higher scores indicating higher levels of emotional lability/negativity.
Time Frame: Baseline and Post-intervention (22 week timepoint)
Population: 2 participants lost to follow up/post-intervention assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 12
score on a scale
  Baseline | 25.33 (3.96)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 22.20 (4.98)

11. Secondary Outcome: Parent Mental Health Symptoms: Anxiety - Hamilton Anxiety Scale (HAM-A)
Description: The Hamilton Anxiety Scale (HAM-A; Hamilton, 1969) is a 14-item self-report measure that assesses physical symptoms of anxiety. Subjects rate the severity of symptoms ranging from 0 (Not present) to 4 (Very Severe). Scores are summed for a total score ranging from 0 to 56, with higher scores indicating higher levels of anxiety.
Time Frame: Baseline and Post-intervention (22 week timepoint)
Population: 2 participants lost to follow up/post intervention assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 12
score on a scale
  Baseline | 19.33 (11.29)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 10.90 (5.78)

12. Secondary Outcome: Parent Mental Health Symptoms: Depression - Patient Health Questionnaire Depression Module (PHQ-9)
Description: The Patient Health Questionnaire - depression module (PHQ-9; Kroenke, Spitzer, & Williams, 2001) is a 9-item self-report questionnaire in which participants rate how often depressive symptoms have bothered them in the past 2 weeks on a scale of 0 (Not at all) to 3 (Nearly every day). Scores are summed for a total score ranging from 0 to 27 with higher scores indicating higher levels of depressed mood.
Time Frame: Baseline and Post-intervention (22 week timepoint)
Population: 2 participants lost to follow up/post-intervention assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 12
score on a scale
  Baseline | 10.42 (6.58)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 4.70 (2.58)

13. Secondary Outcome: Parent Mental Health Symptoms: Substance Craving
Description: The Aggregated Drug Craving Scale (ADCS; Costello et al., 2020) is an adaptation of the Penn Alcohol Craving Scale (PACS; Flannery et al., 1999) aimed at measuring a broad range of substance craving. The measure includes five items that assess intensity, frequency, and duration of craving along with ability to resist substance use if it was available, and it asks responders to give an average craving rating for the past week. The response ranges from 0 to 6 for each item. Responses are summed to provide a total score ranging from 0 to 30, and higher scores indicate greater cravings.
Time Frame: Baseline and Post-intervention (22 week timepoint)
Population: 2 participants lost to follow up/post-intervention assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBT Skills + Parent Training
Number analyzed (Participants) | 12
score on a scale
  Baseline | 9.42 (6.17)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 7.40 (6.69)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | DBT Skills + Parent Training
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT05287178/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT05287178/ICF_002.pdf